CLINICAL TRIAL: NCT00972738
Title: A Multi-Center, Double-blind, Randomized, Parallel-Group Study Investigating the Effect of Montelukast in Patients With Seasonal Allergic Rhinitis-Spring 2001 Study
Brief Title: Montelukast in Seasonal Allergic Rhinitis - Spring 2001 Study (0476-235)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-235; MK0476-235; 2009_658
Record Dates: First submitted 2009-09-04; First posted 2009-09-07 (Estimated); Results first posted 2010-06-16 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): montelukast
  Interventions: Drug: montelukast sodium
- 2 (Active Comparator): loratadine
  Interventions: Drug: Comparator: loratadine
- 3 (Placebo Comparator): placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: montelukast sodium — Montelukast 10-mg tablet orally once daily at bedtime for 2 weeks.
  Arms: 1
Drug: Comparator: loratadine — Loratadine 10-mg tablet orally once daily at bedtime for 2 weeks.
  Arms: 2
Drug: Comparator: Placebo — placebo tablet orally once daily at bedtime for 2 weeks
  Arms: 3

SUMMARY:
This study will assess the treatment effect of montelukast versus placebo over a 2 week period in patients with seasonal allergic rhinitis. Loratadine is included in the study as an active comparator.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a documented history of season allergic rhinitis symptoms that flare up during the study season
* Patient is a nonsmoker
* Patient is in good general health

Exclusion Criteria:

* Patient is hospitalized
* Patient is a woman who is <8 weeks postpartum or is breast-feeding
* Patient has had major surgery in the past 4 weeks
* Patient intends to move or vacation away during the study
* Patient is a current or past abuser of alcohol or illicit drugs

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1214 (Actual)
Dates: Start 2001-04; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] van Adelsberg J, Philip G, LaForce CF, Weinstein SF, Menten J, Malice MP, Reiss TF; Montelukast Spring Rhinitis Investigator Group. Randomized controlled trial evaluating the clinical benefit of montelukast for treating spring seasonal allergic rhinitis. Ann Allergy Asthma Immunol. 2003 Feb;90(2):214-22. doi: 10.1016/S1081-1206(10)62144-8. PMID 12602669

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-two study sites in Canada and the United States.
  Primary Therapy Period: Apr-2001 to Jul-2001.
Pre-assignment Details: Patients who required certain medications as described in the protocol and those who did not meet a minimum predefined level of combined daytime nasal symptoms score during the run-in period were excluded from randomization.
Groups:
- Montelukast 10 mg: Montelukast 10 mg film-coated tablet and loratadine matching-image placebo tablet orally once daily at bedtime for 2 weeks.
- Loratadine 10 mg: Loratadine 10 mg compressed tablet and montelukast matching-image placebo tablet orally once daily at bedtime for 2 weeks.
- Placebo: Montelukast matching-image placebo tablet and loratadine matching-image placebo tablet orally once daily at bedtime for 2 weeks.
Period: Overall Study
Arm/Group | Montelukast 10 mg | Loratadine 10 mg | Placebo
Started | 522 | 171 | 521
Completed | 501 | 165 | 492
Not Completed | 21 | 6 | 29
Not completed — Adverse Event | 7 | 1 | 8
Not completed — Protocol Violation | 2 | 1 | 3
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Lack of Efficacy | 5 | 1 | 11
Not completed — Withdrawal by Subject | 5 | 1 | 4
Not completed — Moved | 0 | 0 | 1
Not completed — Other | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast 10 mg | Loratadine 10 mg | Placebo | Total
Number analyzed (Participants) | 522 | 171 | 521 | 1214
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (13.93) | 34.7 (12.73) | 35.8 (12.61) | 35.5 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 326 | 100 | 338 | 764
  Male | 196 | 71 | 183 | 450
Daytime Eye Symptoms score [Mean (Standard Deviation); unit: Scores on a scale] — Patients were asked to rate each of the 4 eye symptoms of tearing, itchy, red, and puffy eyes daily on a 4-point scale [0 (best) to 3 (worst)]. The average of the 4 individual eye symptoms scores was reported as the Daytime Eye Symptoms Score.
  Scores on a scale | 1.49 (0.77) | 1.48 (0.79) | 1.53 (0.81) | 1.51 (0.79)
Daytime Nasal Symptoms score [Mean (Standard Deviation); unit: Scores on a scale] — Patients were asked to rate each of the 4 nasal symptoms of Congestion, Rhinorrhea, Itching, and Sneezing daily on a 4-point scale [Score 0 (best) to 3 (worst)]. The average of the 4 individual nasal symptoms scores was reported as the Daytime Nasal Symptoms Score.
  Scores on a scale | 2.10 (0.43) | 2.15 (0.45) | 2.14 (0.43) | 2.12 (0.43)
Nighttime Symptoms score [Mean (Standard Deviation); unit: Scores on a scale] — Patients were asked to rate each symptoms of Nasal Congestion Upon Awakening, Difficulty Going to Sleep, and Nighttime Awakenings daily on a 4-point [Scale 0 (best) to 3 (worst)]. The average of the individual symptoms scores was reported as the Nighttime Symptoms Score.
  Scores on a scale | 1.51 (0.65) | 1.49 (0.64) | 1.47 (0.65) | 1.49 (0.65)
Rhinoconjunctivitis Quality-of-Life score [Mean (Standard Deviation); unit: Scores on a scale] — Rhinoconjunctivitis Quality-of-Life score Description (see instructions; limit 350 characters) Self-administered questionnaire which included 28 questions on a 7-point scale [0(best) to 6(worst)] across 7 domains : activity, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotions. Scores for each domain were average, then scores for the 7 domains were averaged for overall score.
  Scores on a scale | 3.22 (1.06) | 3.24 (0.97) | 3.29 (1.01) | 3.25 (1.03)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Daytime Nasal Symptoms Score Over the 2-week Treatment Period
Description: Mean change from baseline in Daytime Nasal Symptoms. Patients were asked to rate each of the 4 nasal symptoms of Congestion, Rhinorrhea, Itching, and Sneezing daily on a 4-point scale [Score 0 (best) to 3 (worst)]. The average of the 4 individual nasal symptoms scores was reported as the Daytime Nasal Symptoms Score.
Time Frame: Baseline and over the 2-week treatment period
Population: The primary efficacy analyses were based on intention-to-treat (all-patients-treated) principle, i.e., all patients who had a baseline and at least one posttreatment measurement were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Montelukast 10 mg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 519 | 170 | 521
Scores on a scale | -0.38 [-0.43 to -0.33] | -0.47 [-0.55 to -0.39] | -0.29 [-0.33 to -0.24]

2. Secondary Outcome: Mean Change From Baseline in Nighttime Symptoms Score Over the 2-week Treatment Period
Description: Mean change from baseline in Nighttime Symptoms Score. Patients were asked to rate each symptoms of Nasal Congestion Upon Awakening, Difficulty Going to Sleep, and Nighttime Awakenings daily on a 4-point [Scale 0 (best) to 3 (worst)]. The average of the individual symptoms scores was reported as the Nighttime Symptoms Score.
Time Frame: Baseline and over the 2-week treatment period
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Montelukast 10 mg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 519 | 170 | 521
Scores on a scale | -0.28 [-0.32 to -0.24] | -0.28 [-0.35 to -0.21] | -0.20 [-0.25 to -0.16]

3. Secondary Outcome: Mean Change From Baseline in Daytime Eye Symptoms Score Over the 2-week Treatment Period
Description: Mean change from baseline in Daytime Eye Symptoms scores. Patients were asked to rate each of the 4 eye symptoms of tearing, itchy, red, and puffy eyes daily on a 4-point scale [0 (best) to 3 (worst)]. The average of the 4 individual eye symptoms scores was reported as the Daytime Eye Symptoms Score.
Time Frame: Baseline and over the 2-week treatment period
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Montelukast 10 mg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 519 | 170 | 521
Scores on a scale | -0.28 [-0.32 to -0.23] | -0.40 [-0.47 to -0.32] | -0.21 [-0.25 to -0.16]

4. Secondary Outcome: Patient's Global Evaluation of Allergic Rhinitis at the End of the 2-week Treatment Period
Description: An evaluation by the patient, administered at the last visit (or upon discontinuation) using a 7-point scale [Score 0 (very much better) to 6 (very much worse)], of the change in symptoms as compared to the beginning of the study.
Time Frame: End of the 2-week treatment period
Population: The primary efficacy analyses were based on the intention-to-treat (all-patients-treated) principle. Since only 1 measurement was obtained during the treatment period, no missing values were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Montelukast 10 mg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 519 | 171 | 517
Scores on a scale | 2.18 [2.05 to 2.31] | 2.19 [1.97 to 2.42] | 2.49 [2.36 to 2.62]

5. Secondary Outcome: Physician's Global Evaluation of Allergic Rhinitis at the End of the 2-week Treatment Period
Description: An evaluation by the physician, administered at the last visit (or upon discontinuation) using a 7-point scale [Score 0 (very much better) to 6 (very much worse)], of the change in symptoms as compared to the beginning of the study.
Time Frame: End of the 2-week treatment period
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Montelukast 10 mg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 521 | 171 | 515
Scores on a scale | 2.18 [2.07 to 2.30] | 2.16 [1.96 to 2.35] | 2.41 [2.29 to 2.52]

6. Secondary Outcome: Mean Change From Baseline in Rhinoconjunctivitis Quality-of-Life Score After the 2-week Treatment Period
Description: Patients completed a validated, self-administered Rhinoconjunctivitis Quality-of-Life Questionnaire, which included 28 questions on a 7-point scale [Score 0 (best) to 6 (worst)], across 7 domains: activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotional. The individual domain scores were calculated as the average values of all scores within a domain, then the scores for the 7 domains were averaged for the overall score.
Time Frame: Baseline and at the end of 2-week treatment period
Population: The primary efficacy analyses were based on the intention-to-treat (all-patients-treated) principle, i.e., all patients who had a baseline and a week 2 measurement were included. No missing values were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Montelukast 10 mg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 518 | 171 | 516
Scores on a scale | -0.90 [-1.00 to -0.81] | -0.98 [-1.15 to -0.81] | -0.66 [-0.76 to -0.56]

ADVERSE EVENTS:
Time Frame: During the two week double-blind treatment period , and up to and including 14 days after the last dose of study therapy.
Arm/Group | Montelukast 10 mg | Loratadine 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/522 | 0/171 | 0/521
Other Adverse Events (participants affected / at risk) | 0/522 | 0/171 | 0/521

LIMITATIONS AND CAVEATS:
In the paper patients who withdrew for worsening allergic rhinitis/conjunctivitis were included under category of discontinued due to lack of efficacy rather than discontinued due to clinical Adverse Events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.